CLINICAL TRIAL: NCT04375423
Title: Mobile Behavioral Ecological Momentary Assessment and Intervention in Rakai, Uganda: A Pilot Study
Brief Title: Mobile Behavioral Ecological Momentary Assessment and Intervention in Rakai, Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Rakai Health Sciences Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00065934
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Ecological Momentary Assessment and Intervention
MeSH Terms: interventions — Ecological Momentary Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): On smartphones, participants in this arm will receive twice daily and weekly prompts to report on behaviors under study and be able to send self-initiated event-contingent reports on behaviors under study. In response to the behaviors they report, they receive messages on their smartphones supporting ongoing healthy behaviors or suggesting alternative behaviors to limit risks. They will complete in-person assessments at enrollment, 30-days and study exit at 90-days.
  Interventions: Behavioral: Ecological momentary assessment and intervention: Behaviorally-dependent messaging; Behavioral: Ecological momentary assessment only
- Control (Active Comparator): On smartphones, participants in this arm will receive twice daily and weekly prompts to report on behaviors under study and be able to send self-initiated event-contingent reports on behaviors under study. They will complete in-person assessments at enrollment, 30-days and study exit at 90-days.
  Interventions: Behavioral: Ecological momentary assessment only

INTERVENTIONS:
Behavioral: Ecological momentary assessment and intervention: Behaviorally-dependent messaging — In response to behavioral data submitted intervention arm participants receive messages on their phones reinforcing healthy behaviors or encouraging alternative behaviors to limit risks
  Arms: Intervention
Behavioral: Ecological momentary assessment only — Participants will receive twice daily and weekly prompts to submit behavioral report data and self-initiate event-contingent behavioral report data submissions

SUMMARY:
Ecological Momentary Assessment and Intervention (EMAI) is an emerging technique for gathering richer and more relevant data through repeated, longitudinal sampling of participants in their natural setting in order to deliver real-time interventions. The main study objective is to conduct a pilot EMAI study in Rakai, Uganda. Secondary objectives are to assess processes, facilitators, and barriers to EMAI. The study will compare behaviors between participants randomized to receive intervention messages and those not receiving messages. To assess EMAI validity and relevance, EMAI-collected behavioral data will be compared with traditional questionnaire-collected data.

After recruitment, participants will be given a smartphone with an application that will collect geospatial coordinates and ask behavioral assessment questions on topics including diet/alcohol, smoking, and sexual behaviors. Participants will have training on the phone and application, demonstrating proficiency with the EMAI interface prior to study start.

Days 1-30, Baseline Behaviors: Participants will complete assessment questions to establish baseline behaviors. This will include twice-daily and weekly behavioral report prompts and participant-initiated event-contingent behavioral reports. After the initial 30 day period, participants will return to the study office to complete a short questionnaire and to be randomized to the second phase of follow-up.

Days 31-90, Randomized Evaluation: Participants will be randomized in a 1:1 ratio to either continue assessment questions only (control arm) or to also begin receiving intervention messages (intervention arm) in response to reported behaviors. Messages will encourage positive behaviors and suggest alternatives to negative behaviors (e.g. "Eating a mixed diet (meats and vegetables) is a healthy way to go."). At 90 days of follow-up, participants will return to the study office to complete a brief questionnaire on behaviors and smartphone experiences.

Study hypotheses are as follows: EMAI can be successfully implemented in Uganda, and participants receiving intervention messaging will have improved self-reported health behaviors compared to controls; EMAI will be feasible and acceptable by this population; and, EMAI-collected data will correlate with traditional questionnaire-collected data.

Outcomes will be assessed using descriptive statistics, multivariate regression and analysis of themes in patient EMAI experience and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* literate
* current Rakai Community Cohort Study participant

We will purposely recruit a sample that has a broad range of participant characteristics in our study to optimize diversity of responses and increase study generalizability. Specific variables for which we will target sampling include: gender (~50% female), age (at least 20% among age groups 18-25, 26-35, >50), and occupation (at least 20% traders and farmers).

Exclusion Criteria:

* Participants without a listed phone number in the Rakai Community Cohort Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change in health behavior according to EMAI self-report | Daily, comparing baseline (days 1-30) to follow up (days 31-90), up to a total 90 days
  change in the proportion of days when participant reports 'yes' to behavior over total days behavior measured, comparing baseline to follow-up in self-reported: alcohol consumption, fruit and vegetable consumption; cigarette smoking, and sex with a non-longterm or non-marital partner

CONTACTS AND LOCATIONS:
Overall Officials: Larry Chang, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beres LK, Mbabali I, Anok A, Katabalwa C, Mulamba J, Thomas AG, Bugos E, Nakigozi G, Grabowski MK, Chang LW. Mobile Ecological Momentary Assessment and Intervention and Health Behavior Change Among Adults in Rakai, Uganda: Pilot Randomized Controlled Trial. JMIR Form Res. 2021 Jul 20;5(7):e22693. doi: 10.2196/22693. PMID 34283027

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/23/NCT04375423/Prot_SAP_000.pdf